CLINICAL TRIAL: NCT02478528
Title: Study of Effects of Light on the Vigilance and Cognitive Performance Following a Night Without Sleep
Acronym: LUMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6191
Record Dates: First submitted 2015-01-26; First posted 2015-06-23 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Device: Energy-Light lamp; Device: Luminettes lamp; Other: control condition

INTERVENTIONS:
Device: Energy-Light lamp — Exposure of the subject, at 5am, to the light source of Energy-Light lamp (Philips)
Device: Luminettes lamp — Exposure of the subject, at 5am, to the light source of Luminettes lamp (Lucimed)
Other: control condition — No exposure of the subject to any light sources (control condition)

SUMMARY:
Sleep disorders are a major public health issue, affecting 1 in 6 French. The medical impact at the individual level but also social and economic level (loss of productivity, morbidity, mortality) emphasize the need for one hand, to improve the investigators' understanding of these disorders in order to develop appropriate therapeutic tools and on the other hand, to increase the investigators' support abilities of patients with these disorders.

The investigators' team of unity sleep from Strasbourg University Hospitals, in collaboration with the UPR 3212 CNRS team, is working on the development and adjustment of new concepts and tools to compensate the investigators' sleep debt in order to apply them to patients with sleep disorders and persons who face with sleep restriction.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Age from 18 to 40 years
* With a Body Mass Index (BMI) between 17 and 30 kg m-2
* Healthy volunteer determined by clinical examination and psychological interview
* Agreeing to abstain from caffeine, nicotine, alcohol, psychotropic drugs, cannabis or other drugs, the week before the start of Stage 2 of the study until the end of the study
* Dated and signed informed consent
* Subjet affiliated to a social security scheme
* Subject has been informed about the results of the medical examination

Exclusion Criteria:

* Participation in other clinical trials in the month preceding the inclusion
* Shift work in the year before inclusion
* Cons-indications to the use of the medical device
* Ocular disease
* Unable to give informations to the subject (subject in an emergency situation, difficulties in understanding, ...)
* Subjet under judicial protection
* Subject under guardianship or curatorship
* pregnancy
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Analysis of the perception of fatigue | Compare during the 3 sessions : energy-light lamp, luminettes lamp and control condition
  Karolinska Sleepiness Scale 3 sessions :
Analysis of the circadian variation of melatonin and cortisol secretion | Compare during the 3 sessions : energy-light lamp, luminettes lamp and control condition
  cortisol and melatonin dosage

SECONDARY OUTCOMES:
Cognitive performance | Compare during the 3 sessions : energy-light lamp, luminettes lamp and control condition
  neurobehavioral tests

CONTACTS AND LOCATIONS:
Locations (1):
- Unité du Sommeil - Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Result] Comtet H, Geoffroy PA, Kobayashi Frisk M, Hubbard J, Robin-Choteau L, Calvel L, Hugueny L, Viola AU, Bourgin P. Light therapy with boxes or glasses to counteract effects of acute sleep deprivation. Sci Rep. 2019 Dec 2;9(1):18073. doi: 10.1038/s41598-019-54311-x. PMID 31792259